CLINICAL TRIAL: NCT02059993
Title: The Effects of Obstructive Sleep Apnea and Its Intervention on Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SF2009-2012
Record Dates: First submitted 2014-02-09; First posted 2014-02-11 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Hypertension; Metabolic Disorder
Keywords: continuous positive airway pressure; hypertension; coronary heart disease; metabolic disorder; obstructive sleep apnea
MeSH Terms: conditions — Hypertension; Metabolic Diseases; Coronary Disease; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- continuous positive airway pressure (Other): mean continuous positive airway pressure use was at least 4 hours per night; continuous positive airway pressure group received fixed-level continuous positive airway pressure titration using an automated pressure
  Interventions: Device: continuous positive airway pressure
- Control (No Intervention): The control subjects received standardised anti-hypertension medications according to the current guildline.

INTERVENTIONS:
Device: continuous positive airway pressure — mean continuous positive airway pressure use was at least 4 hours per night;continuous positive airway pressure group received fixed-level continuous positive airway pressure titration using an automated pressure
  Arms: continuous positive airway pressure

SUMMARY:
Obstructive sleep apnea(OSA) is an important identifiable cause of hypertension. Previous study has suggested that OSA significantly increases cardiovascular morbidity and mortality, especially in patients with pre-existing cardiovascular disease.The standardized treatment of moderate/severe OSA is continuous positive airway pressure (CPAP). Most of short-term trials indicated that CPAP treatment reduced BP in patients with OSA. But relevant studies have a relative short duration with only but few more than one year. In our opinion, they are not sufficient to detect the real effect of CPAP on reduction in BP. Besides, the impact of OSA on metabolic disorder is still unclear.We hypothesized that long-term CPAP treatment could reduce blood pressure and improve metabolic disorder in patients with coronary heart disease (CHD)and OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder characterized by repetitive partial (hypopnea) or complete (apnea) occlusion of the upper airway during sleep caused by collapse of the pharyngeal airway, resulting in sleep fragmentation and oxyhemoglobin desaturation. Kiely and colleague's study showed that over 20% of hypertensive patients exhibit OSA, whereas prevalence of hypertension in the setting of OSA exceeds 50%. One study confirmed that OSA is an important identifiable cause of hypertension. OSA is considered as one of the most common risk factors of resistant hypertension. Previous study has suggested that OSA significantly increases cardiovascular morbidity and mortality, especially in patients with pre-existing cardiovascular disease. Several studies confirmed that CPAP reduced systolic blood pressure (SBP) and diastolic blood pressure (DBP) in patients with OSA. Additionally, some papers reported that there was a protective effect of CPAP therapy against death from cardiovascular disease in patients with severe OSA. Other researches regarding the antihypertensive effect of CPAP therapy, however, showed that CPAP had no antihypertensive effect. But relevant studies have a relative short duration with only but few more than one year. In our opinion, they are not sufficient to detect the real effect of CPAP on reduction in BP. According to our knowledge, there is no report about long-term effect of CPAP on BP in hypertensive patients with coronary revascularization (CRV) and OSA under conventional antihypertensive medications. Therefore, we conducted a long-term, prospective controlled study to investigate the effects of CPAP on BP, metabolic disorder, clinical symptoms, cardiovascular and cerebrovascular events in patients with CHD and OSA on conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* men and women, aged 45 to 75 years old
* verified diagnosis of hypertension by medical history or receiving antihypertensive drugs
* established diagnosis of CHD
* at least 3-month optimal treatment for hypertension
* moderate or severe OSA

Exclusion Criteria:

* if they had secondary hypertension
* central sleep apneas
* history of significant chronic renal, or hepatic failure or severe pulmonary disease
* diagnosed with malignant cancer with a life expectancy of less than 2years
* regular use of medications that can affect BP(including corticosteroids or sedative drugs)
* severe psychiatric disease
* sustained excessive alcohol use
* current use of CPAP treatment for OSA or pharyngeal surgery for OSA
* New York Heart Association Class III-IV degree
* declined to participate or were unable to give informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD，PhD, Study Chair — Fuwai Hospital, National Center for Cardiovascular Diseases

REFERENCES:
- [Derived] Huang Z, Liu Z, Luo Q, Zhao Q, Zhao Z, Ma X, Liu W, Yang D. Long-term effects of continuous positive airway pressure on blood pressure and prognosis in hypertensive patients with coronary heart disease and obstructive sleep apnea: a randomized controlled trial. Am J Hypertens. 2015 Mar;28(3):300-6. doi: 10.1093/ajh/hpu147. Epub 2014 Aug 14. PMID 25125635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited consecutive patients from outpatient and inpatient departments of Fuwai Hospital from January 2009 to June 2012. Patients were randomly assigned to either continuous positive airway pressure (CPAP) group or no CPAP therapy (control).
Pre-assignment Details: A total of 243 patients were screened between January 2009 and June 2012. Out of 97 (39.9%) patients diagnosed with obstructive sleep apnea (OSA), 5 subjects declined to participate in the study, and 9 subjects were excluded because of the following: apnea-hypopnea index (AHI) <15 (n = 8 patients) and severe heart failure (n = 1 patient).
Groups:
- Continuous Positive Airway Pressure(CPAP) Group: The continuous positive airway pressure group received fixed-level continuous positive airway pressure titration using an automated pressure and the the cardiovascular drugs based on the guidelines.
- Control: The controls only received the cardiovascular drugs based on the guidelines but without continuous positive airway pressure machine.
Period: Overall Study
Arm/Group | Continuous Positive Airway Pressure(CPAP) Group | Control
Started | 42 | 41
Completed | 40 | 37
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Population: A total of 243 patients were screened between January 2009 and June 2012. Out of 97 (39.9%) patients diagnosed with OSA, 5 subjects declined to participate in the study, and 9 subjects were excluded because of the following: AHI <15 (n = 8 patients) and severe heart failure (n = 1 patient).
Groups:
- Continuous Positive Airway Pressure(CPAP) Group: The CPAP group received fixed-level CPAP titration using an automated pressure setting device for one night. The optimal CPAP pressure for each patient in the CPAP group was set at the minimum pressure required to abolish snoring, obstructive respiratory events, and airflow limitation for 95% of the night.
- Control: The control group received the standardized antihypertensive medications but without receiving CPAP machine.
- Total: Total of all reporting groups
Arm/Group | Continuous Positive Airway Pressure(CPAP) Group | Control | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (6.8) | 62.7 (6.7) | 62.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 30 | 31 | 61
Region of Enrollment [Number; unit: participants]
  China | 42 | 41 | 83
morning systolic and diastolic BP (mmHg) [Mean (Standard Deviation); unit: mm Hg] — The morning BP was measured with a mercury sphygmomanometer by an experienced physician unaware of the patient's group assignment,which was the main end point.
  mm Hg
    systolic BP | 146 (8) | 148 (11) | 147 (9)
    diastolic BP | 83 (7) | 83 (8) | 83 (7)

OUTCOME MEASURES:

1. Primary Outcome: Change of Daytime Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Pre-treatment and Post-treatment
Time Frame: baseline and follow-up at 36 months
Population: 4 participants withdrew before the end of study. Two subjects were lost to follow-up in the control group, and 4 patients (all of them had no SCCE) with very poor CPAP compliance were also excluded.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Continuous Positive Airway Pressure(CPAP) Group: The subjects who received CPAP treatment and standardized medicine.
- Control: The patients who use standardized drugs without CPAP machine.
Arm/Group | Continuous Positive Airway Pressure(CPAP) Group | Control
Number analyzed (Participants) | 36 | 37
mm Hg
  Change of SBP | -8 (11) | -3 (6)
  Change of DBP | -4 (11) | -3 (11)
Statistical Analysis 1: Comparison: Continuous Positive Airway Pressure(CPAP) Group vs Control; The sample size was calculated to assess a minimum reduction of 5 ± 5 mm Hg in systolic BPafter CPAP treatment, assuming an alpha error of 5% and a statistical power of 80%; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 10

2. Secondary Outcome: Change in Epworth Sleepiness Scale (ESS)
Description: The epworth sleepiness scale（ESS） measures a person's general level of daytime sleepiness, or their average sleep propensity in daily life (ASP). It is a simple questionnaire based on retrospective reports of the likelihood of dozing off or falling asleep in a variety of different situations. The ESS is the most commonly used method for measuring a person's ASP.The ESS ranges from 0-24, higher scores indicate more severe daytime sleepiness.
Time Frame: baseline，end of study ( up to 54 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous Positive Airway Pressure(CPAP) Group | Control
Number analyzed (Participants) | 36 | 37
score on a scale | 7.0 (3.4) | 3.7 (2.3)
Statistical Analysis 1: Comparison: Continuous Positive Airway Pressure(CPAP) Group vs Control; Test type: Other; p = 0.001, t-test, 2 sided

3. Other Pre Specified Outcome: Cardiovascular and Cerebrovascular Events
Time Frame: Baseline, 1 month, 3 month, 6 month, 12 month, 18 month, 24 month, 30 month, 36 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Description: SCCEs included new-onset acute myocardial infarction (AMI), hospitalization for heart failure, need for repeated coronary revascularization, stroke, and death associated with cardiovascular and cerebrovascular disease.
Groups:
- Continuous Positive Airway Pressure(CPAP) Group: The CPAP group received fixed-level CPAP titration using an automated pressure setting device for 1 night. The optimal CPAP pressure for each patient in the CPAP group was set at the minimum pressure required to abolish snoring, obstructive respiratory events, and airflow limitation for 95% of the night.
Arm/Group | Continuous Positive Airway Pressure(CPAP) Group | Control
Serious Adverse Events (participants affected / at risk) | 1/42 | 5/41
Other Adverse Events (participants affected / at risk) | 0/42 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Positive Airway Pressure(CPAP) Group (N=42) | Control (N=41)
acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
heart failure (Cardiac disorders) | 1 (1) | 0 (0)
stroke (Nervous system disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
First, the sample size was relatively small. Second, this was a nondouble-blind study. Third, we did not use 24-hour ambulatory BP to monitor changes in BP and could not evaluate the nighttime BP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No